CLINICAL TRIAL: NCT07045727
Title: Prehabilitation in Patients With Multiple Myeloma Receiving CAR-T Therapy
Brief Title: Prehabilitation With Aerobic and Resistance Exercise for Improving Physical Fitness and Quality of Life Outcomes in Older Patients Undergoing CAR-T Therapy for Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-001845; NCI-2025-04165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-001845 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Accelerometry; Exercise; Specimen Handling; Interviews as Topic; Exercise Test; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (aerobic and resistance training) (Experimental): Patients receive a personalized exercise plan and use the Connected mHealth app to participate in aerobic and resistance training, according to exercise guidelines and their personalized plan, for 6 weeks. Patients also receive health coaching check-in calls weekly for 6 weeks. Patients also undergo collection of blood and urine samples throughout the study.
  Interventions: Procedure: Accelerometry; Other: Aerobic Exercise; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Exercise Counseling; Other: Internet-Based Intervention; Other: Interview; Other: Physical Performance Testing; Other: Resistance Training; Other: Survey Administration; Procedure: Tailored Intervention

INTERVENTIONS:
Procedure: Accelerometry — Ancillary studies
Other: Aerobic Exercise — Participate in aerobic training program
  Other Names: Aerobic Activity
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Other: Exercise Counseling — Receive health coaching check-in calls
Other: Internet-Based Intervention — Use Connected mHealth app
Other: Interview — Ancillary studies
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Resistance Training — Participate in resistance training program
  Other Names: Strength Training
Other: Survey Administration — Ancillary studies
Procedure: Tailored Intervention — Receive personalized exercise plan

SUMMARY:
This clinical trial evaluates whether prehabilitation with aerobic and resistance exercise improves physical fitness and quality of life outcomes in older patients planning to undergo chimeric antigen receptor (CAR)-T therapy for multiple myeloma that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). CAR-T therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. Large numbers of the CAR-T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. While CAR-T therapy is commonly used to treat multiple myeloma, it can result in toxicities that lead to hospitalization, nerve and muscle impairment, and decreased physical function. Prehabilitation programs use targeted interventions to improve functional status prior to medical or surgical treatments. In this study, patients participate in personalized aerobic and resistance prehabilitation activities in the weeks leading up to their CAR-T infusion. This program may improve physical fitness and quality of life, both prior to and after CAR-T infusion, in older patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma diagnosis
* Females and males ≥ 60 years of age
* Eastern Cooperative Oncology Group (ECOG) score of < 3
* Scheduled for a CAR T therapy transfusion
* Apheresis date at least 7 days prior to date of enrollment
* Primary hematologist attending physician clearance for exercise

Exclusion Criteria:

* Females or males < 60 years of age
* Any hematological cancer other than multiple myeloma
* Evidence of an absolute contraindication [e.g., heart insufficiency > New York Heart Association (NYHA) III or uncertain arrhythmia; uncontrolled hypertension; reduced standing or walking ability for exercise]
* Other comorbidities that preclude participation in the exercise as deemed by physical therapist or physical medicine and rehabilitation (PM&R) physician
* Active infections, active bleeding disorders, and cytopenias at risk for further adverse events deemed by hematologist-oncologist

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | Up to 1 year
  Enrollment rate will be evaluated as the number of patients eligible versus the number of patients enrolled.
Retention rate | Up to 30 days post-chimeric antigen receptor (CAR)-T infusion
  Retention rate will be evaluated as the proportion of enrolled patients who complete assessments at visit 2 (at 2 days prior to CAR-T infusion) and visit 3 (30 days post-CAR-T infusion).
Program completion | Up to 30 days post-CAR-T infusion
  Will be evaluated according to the completion of weekly phone calls, the frequency, intensity, and duration of exercise engagement, and accelerometer summary outcomes. The program will be considered feasible if there is > 70% program completion, based on weekly phone calls.
Incidence of adverse events | Up to 30 days post-CAR-T infusion
  The program will be considered feasible if there are no serious adverse events due to the intervention.
Patient satisfaction | Up to 30 days post-CAR-T infusion
  Patient satisfaction will be determined using post-program satisfaction phone interviews. Qualitative interviews will be analyzed using thematic analysis.
Change in muscle strength | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  Assessed as grip strength, as measured (in kg) by maximal force generated by forearm muscles using calibrated handheld dynamometer
Change in muscle mass | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  Assessed via SOZO by ImpediMed [bioimpedance spectroscopy (BIS)] and Positron Emission Tomography (PET) Computed Tomography (CT) CT scan images, obtained as part of the patient's usual care.
Change in physical performance | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  Assessed via short physical performance test (approximately 90 minutes) followed by wearing an activity monitor (Actigraph) for 7 days following each of 3 in-person physical assessments. Participants receive a postage-paid envelope to return the monitor after wearing it.
Change in quality of life - EORTC QLQ-C30 | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  Assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30, a 30-item questionnaire where 28 questions are answered on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, and 4= very much) and 2 two questions are answered on a scale of 1-7 (1= very poor and 7=excellent). Higher summary scores indicate better health related quality of life.
Change in physical activity - monitor | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  Assessed using Polar heart rate monitor with data collected through the Connected mHealth app.
Change in physical activity - RPE Scale | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  Assessed using patient self-reported Rate of Perceived Exertion (RPE) scale score within the Connected mHealth app after exercise: 1=very light activity; 2-3=light activity; 4-5=moderate activity; 7-8=vigorous activity; 9=very hard activity; and 10=maximal effort.
Changes in frailty status - IMWG-FI | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  Assessed using International Myeloma Working Group (IMWG) Frailty Index (FI) scores. The IMWG-FI assigns scores based on age, comorbidities, and the ability to perform activities of daily living (ADL) and instrumental activities of daily living (IADL). Patients are categorized as follows: Fit: Score of 0; Intermediate-fit: Score of 1; Frail: Score of 2 or higher.
Changes in frailty status - FP | Baseline (prior to the intervention; Visit 1); Post-intervention (two days prior to CAR-T infusion; Visit 2), Follow-up (Day 30 post CAR-T; Visit 3)
  The Fried frailty phenotype (FP) defines frailty as the presence of three or more of the following: unintentional weight loss ≥10 lb in previous year; self-reported exhaustion; weakness measured by grip strength; slow walking speed ;and low physical activity (less than 3 days of physical activity per week defined by the Department of Health Services & Human Services). The presence of: 1) ≥3 criteria indicates frail status, 2) 1 or 2 criteria indicates intermediate or pre-frail status, and 3) 0 criteria indicates robust status.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine H. Abdallah, MD, Principal Investigator — Mayo Clinic; Diane K. Ehlers, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials